CLINICAL TRIAL: NCT00481325
Title: A Multicenter, Randomized, Double-Blind, Placebo and Escitalopram Controlled Trial of the Safety and Efficacy of Pexacerfont (BMS-562086) in the Treatment of Outpatients With Generalized Anxiety Disorder
Brief Title: Study of Pexacerfont (BMS-562086) in the Treatment of Outpatients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN148-015
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — pexacerfont; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Experimental)
  Interventions: Drug: pexacerfont
- A2 (Active Comparator)
  Interventions: Drug: escitalopram
- A3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pexacerfont — Tablets & Capsules, Oral, 300mg loading dose then 100 mg, once daily, 1 week loading dose then 8 weeks
  Other Names: (BMS-562086)
  Arms: A1
Drug: escitalopram — Tablets & Capsules, Oral, 10-20mg, once daily, 1 week loading dose then 8 weeks
  Arms: A2
Drug: placebo — Tablets & Capsules, Oral, 0 mg, once daily, 1 week loading dose then 8 weeks
  Arms: A3

SUMMARY:
The purpose of this study is to learn about the safety and efficacy of pexacerfont in outpatients diagnosed with Generalized Anxiety Disorder

ELIGIBILITY:
Inclusion Criteria:

* Outpatient women ages 18-65 meeting Diagnostic and Statistical Manual of Mental Disorders Manual, Fourth Edition, Text Revision (DSM-IV TR) criteria for Generalized Anxiety Disorder (GAD), either moderate or severe (300.02)

Exclusion Criteria:

* Males
* Patients who report a history of inadequate response to three or more adequate trials of any selective Serotonin reuptake inhibitors (SSRIs) for GAD within the last three years

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 8 on the Site-Rated Hamilton Anxiety Rating Scale (total score) | Week 8

SECONDARY OUTCOMES:
Mean change from baseline to Week 8 on the Sheehan Disability Scale (SDS) Total Score | Week 8
Mean change from baseline to Week 8 on the Gastrointestinal Symptom Index Total Score | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (51):
- United States (51):
  - Pivotal Research Centers, Mesa, Arizona
  - Pacific Clinical Research Medical Group, Burbank, California
  - Us Clinical Research Centers, Llc, Costa Mesa, California
  - Pacific Institute For Medical Research, Inc., Los Angeles, California
  - Affiliated Research Institute, San Diego, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Radiant Research, Inc., Denver, Colorado
  - University Of Connecticut Health Center, Farmington, Connecticut
  - Comprehensive Psychiatric Care, Pc, Norwich, Connecticut
  - Meridien Research, Brooksville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Comprehensive Neuroscience, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Carman Research, Smyrna, Georgia
  - Indiana University School Of Medicine, Indianapolis, Indiana
  - Alpine Clinic, Lafayette, Indiana
  - Cientifica, Inc. At Prairie View Inc., Newton, Kansas
  - Ctt, Inc., Prairie Village, Kansas
  - J. Gary Booker, Md, Apmc, Shreveport, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Capital Clinical Research Associates, Rockville, Maryland
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - Regions Hospital, Saint Paul, Minnesota
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Bioscience Research, Llc, New York, New York
  - Fieve Clinical Services, Inc., New York, New York
  - Social Psychiatry Research Institute, New York, New York
  - Behavioral Medical Research Of Staten Island, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - North Carolina Neuropsychiatry, Pa, Charlotte, North Carolina
  - Medark Clinical Research, Morganton, North Carolina
  - Psychiatry And Clinical Research, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Ips Research Company, Oklahoma City, Oklahoma
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Center For Clinical Investigations, Inc. (Occi, Inc), Salem, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina
  - Carolina Clinical Research Services, Llc, Columbia, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Futuresearch Trials, Austin, Texas
  - Futuresearch Trials Of Dallas, Dallas, Texas
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - Medlabs Research Of Houston, Inc., Houston, Texas
  - Red Oak Psychiatry Associates, Pa, Houston, Texas
  - Dominion Clinical Research, Midlothian, Virginia
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin

REFERENCES:
- [Derived] Coric V, Feldman HH, Oren DA, Shekhar A, Pultz J, Dockens RC, Wu X, Gentile KA, Huang SP, Emison E, Delmonte T, D'Souza BB, Zimbroff DL, Grebb JA, Goddard AW, Stock EG. Multicenter, randomized, double-blind, active comparator and placebo-controlled trial of a corticotropin-releasing factor receptor-1 antagonist in generalized anxiety disorder. Depress Anxiety. 2010 May;27(5):417-25. doi: 10.1002/da.20695. PMID 20455246